CLINICAL TRIAL: NCT01690052
Title: Efficacy of Cevimeline vs. Pilocarpine in the Secretion of Saliva
Brief Title: Efficacy of Cevimeline Versus Pilocarpine in the Secretion of Saliva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Joel Thompson, PhD, PRS administrator, University of Kentucky
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 9999
Record Dates: First submitted 2011-04-06; First posted 2012-09-21 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Dry Mouth
Keywords: dry mouth
MeSH Terms: conditions — Xerostomia | interventions — cevimeline; Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cevimeline (Active Comparator): Cevimeline vs Pilocarpine
  Interventions: Drug: Cevimeline
- Pilocarpine (Active Comparator): Pilocarpine vs. Cevimeline
  Interventions: Drug: Pilocarpine

INTERVENTIONS:
Drug: Cevimeline — Cevimlenine Vs Pilocarpine, cross over design. Two sequences were evaluated "cevimeline first, then pilocarpine" and "pilocarpine first, then cevimeline". Each sequence was evaluated for 4 weeks with one week "washout" period in between both sequences. 15 patients were randomly assigned to a specific sequence by a research pharmacist independent from the study authors. The patients received 30mg of cevimeline three times a day and pilocarpine 5mg three times a day.
  Arms: Cevimeline
Drug: Pilocarpine — Cevimlenine Vs Pilocarpine, cross over design, 4 weeks, one week wash out
  Arms: Pilocarpine

SUMMARY:
The main objectives were: 1) To determine the efficacy of both cevimeline and pilocarpine in the secretion of saliva in patients with xerostomia, and 2) To compare the side-effects between the treatment for xerostomia with cevimeline and with pilocarpine.

DETAILED DESCRIPTION:
Pilocarpine is a cholinergic agonist with predominant muscarinic action.As such, it acts at muscarinic-cholinergic receptors found throughout the body and promotes fluid secretion. Due to this, one of the main side-effects of pilocarpine is an increased amount of sweating. Thus, not only are the salivary glands stimulated, but all of the body's exocrine glands' production is heightened. On the other hand, cevimeline is a drug with a high affinity for specific muscarinic receptors (M3) located on lachrymal and salivary gland epithelium. At least in theory, cevimeline will produce less side effects compared with pilocarpine because of the higher affinity for the muscarinic receptors located in the salivary glands. A limited number of human clinical trials in the efficacy of cevimeline and pilocarpine to increase the production of saliva and the side effects have been performed with no conclusive results.

The main purposes of this study were to determine the efficacy of cevimeline and pilocarpine in the secretion of saliva in patients with xerostomia, and to compare the side-effects between these two medications.

ELIGIBILITY:
Potential candidates with the diagnosis of moderate-severe xerostomia were identified from the Oral Medicine Clinic at the University Of Kentucky College Of Dentistry, or self referrals in response to IRB approved study announcements. Enrollment required no clinical evidence of oral lesions, subjective perception of dry mouth and less than 2 mL of saliva collected in 5 minutes without stimulation. Exclusion criteria included patients with non controlled chronic obstructive pulmonary disease (COPD), depression, asthma, cardiac arrhythmias, glaucoma, and the current use of any medication with interactions with cevimeline and pilocarpine.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Thompson, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Orofacial Pain Center College of Dentistry, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Salivary Gland Dysfunction Clinic at the U. of K. A cross-over double-blind randomized trial was designed. Two arms were assembled. First arm the SEQUENCE was cevimeline(C) then pilocarpine(P), and for the second the SEQUENCE was P then C. Each participant received the drug for 4 weeks with 1 week washout period.
Pre-assignment Details: The total number of patients screened for the study was 28. Of 28 patients, 15 met the inclusion criteria
Groups:
- Cevimeline First, Then Pilocarpine: Cevimeline First then Pilocarpine: Cevimeline (30mg three times a day) for 4 weeks (First intervention period) and then pilocarpine (5 mg three times a day) for 4 weeks (second intervention period). In between first and second intervention period, participants had a washout period for one week.
- Pilocarpine First, Then Cevimeline: Pilocarpine First then Cevimeline: Pilocarpine (5 mg three times a day) for 4 weeks (first intervention period) and then Cevimeline (30mg three times a day) for 4 weeks (second intervention period). In between first and second intervention period, participants had a washout period for one week.
Period: FIRST INTERVENTION: 4 WEEKS
Arm/Group | Cevimeline First, Then Pilocarpine | Pilocarpine First, Then Cevimeline
Started | 7 | 8
Completed | 6 | 6
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Period: Washout Period of 1 Week
Arm/Group | Cevimeline First, Then Pilocarpine | Pilocarpine First, Then Cevimeline
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: SECOND INTERVENTION: 4 WEEKS
Arm/Group | Cevimeline First, Then Pilocarpine | Pilocarpine First, Then Cevimeline
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Two interventions were assembled:
  For the first intervention, the SEQUENCE was cevimeline (30mg three times a day) for 4 weeks and then Pilocarpine (5 mg three times a day) for 4 weeks, after the first sequence, the participants had a washout period for one week.
  For the second intervention, the SEQUENCE was Pilocarpine (5mg three times a day) or 4 weeks and then Cevimeline (30 mg three times a day) for 4 weeks, after the first sequence, the participants had a washout period for one week.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Saliva Production in ml.
Description: The primary outcome measure was the change of stimulated and non-stimulated saliva in ml from the baseline record.
  At each appointment (weekly), participants will provide 2 saliva samples to measure their current salivary output. The first measurement will be obtained by having the patient spit as much as he or she could into a cup for five minutes. The amount of saliva in ml will be recorded.
  The second measurement will be obtained in a similar manner with the addition of having the patient chew on a block of unflavored wax. Patients will complete weekly questionnaires to help determine which side-effects they experience as they take the medications.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Cevimeline: Cevimeline 30mg administered three times a day in first intervention period or second intervention period for 4 weeks.
- Pilocarpine: Pilocarpine 5 mg administered three times a day in either first intervention period or second intervention period
Arm/Group | Cevimeline | Pilocarpine
Number analyzed (Participants) | 12 | 12
ml
  Unstimulated Saliva | 1.41 (0.5) | 3.93 (0.5)
  Stimulated Saliva | 5.31 (0.5) | 10.34 (0.5)
Statistical Analysis 1: Comparison: Cevimeline vs Pilocarpine; Test type: Superiority or Other; p = 0.05, ANOVA; The p-value is calculated from the ANOVA

2. Other Pre Specified Outcome: Adverse Events
Description: Adverse events related to the combination and order of study medication will be measured
Time Frame: four weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse events are reported per intervention (4 weeks with each medication)
Description: No adverse events were presented in any of the intervention sequences
Groups:
- Cevimeline Then Pilocarpine (Intervention 1): Cevimeline then pilocarpine One week washout period
- Pilocarpine Then Cevimeline (Intervention 2): Pilocarpine then cevimeline One week washout period
Arm/Group | Cevimeline Then Pilocarpine (Intervention 1) | Pilocarpine Then Cevimeline (Intervention 2)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
There are limitations that affected this study. This is a pilot study with a relative low number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No